CLINICAL TRIAL: NCT03892291
Title: Objective Dual-task Turning Measures for Return-to-duty Assessments
Acronym: reTURN
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Courage Kenny Research Center (Unknown); University of Utah (Other); Fort Sam Houston (Unknown); Warrior Recovery Center (Unknown); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie King, Associate Professor, Oregon Health and Science University
Other Study IDs: 18749; W81XWH1820049 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-03-13; First posted 2019-03-27 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Mild Traumatic Brain Injury; Gait; Balance; Veterans; Mobility
Keywords: mild traumatic brain injury; dual-task; veterans; mobility
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Civilian mTBI: Civilians with persistent symptoms from mTBI
- Civilian Control: Civilian healthy controls
- Active Duty Control: Active duty service member healthy controls
- Active Duty mTBI: Active duty service members with persistent symptoms from mTBI who are referred for physical therapy due to their symptoms

SUMMARY:
The overall objective is to evaluate objective dual-task turning measures for use as rehabilitative outcomes and as tools for return-to-duty assessments in individuals with mild traumatic brain injury (mTBI).This project consists of three goals examining the I) Diagnostic Accuracy, II) Predictive Capacity, and III) Responsiveness to Intervention of dual task turning measures in individuals with mTBI.

The investigators hypothesize that objective measures of dual-task turning will have high diagnostic accuracy, predictive capacity, and responsiveness to intervention in people with mTBI.

DETAILED DESCRIPTION:
The purpose of this project is to expand the investigators' prior preliminary work on wearable sensors to evaluate objective dual-task turning measures for use as rehabilitative outcomes and as tools for objective return-to-duty assessments following mild traumatic brain injury (mTBI). The investigators will assess the diagnostic accuracy, predictive capacity, and responsiveness to intervention of measures obtained from clinically feasible, dual-task turning tasks in an effort to evaluate the utility of turning measures for clinical return-to-duty decisions.

This study is divided into two phases. For phase one, participants will be recruited from the general populations surrounding four sites (Oregon Health & Science University, the University of Utah, Courage Kenny Research Center, and Fort Sam Houston), including active duty service members at Fort Sam Houston. For phase two, participants will be recruited from active duty service members referred to military medical treatment facilities (Warrior Recovery Center, Madigan Army Medical Center) for vestibular rehabilitation following mTBI.

Phase One: Fifty civilian individuals with mTBI, 50 healthy control individuals, and 40 healthy control active duty service members will be recruited for phase one. Participants will complete a battery of clinical, neuropsychological, and balance tests, including three clinically feasible turning tasks while wearing inertial sensors. The investigators will evaluate the capability of objective, dual-task turning measures to discriminate between healthy controls and people with chronic mTBI, determine clinically relevant measures of dual-task turning based on clinometric properties (e.g., minimum detectable change), and determine whether active-duty SMs perform dual-task turning tasks differently than civilians, assess the capacity of dual-task turning measures to predict performance in a civilian-relevant task, and assess the capacity of dual-task turning measures to predict performance in a military-relevant task.

Phase Two: Forty active-duty service members with mTBI referred to vestibular rehabilitation at the Warrior Recovery Center or Madigan Army Medical Center will be recruited for phase two. Participants will complete a selected turning task from phase one at the beginning and end of the treatment. The investigators will determine the clinically important difference of turning outcomes and compare the effect of rehabilitation to the minimum detectable change for each outcome.

ELIGIBILITY:
Inclusion criteria.

Participants may be active duty (at FSH), Veterans or non-Veterans or a civilian and must:

1. have a diagnosis of mTBI based upon VA/DoD criteria
2. be between 18-50 years-old,
3. be outside of the acute stage (> 3 weeks post-concussion) according to the VA/DoD clinical practice guidelines but within 3 years of their most recent mTBI and still reporting symptoms.

Exclusion criteria.

Participants must not:

1. have had or currently have any other injury, medical, or neurological illness that could potentially explain balance deficits (e.g., central or peripheral nervous system disease, stroke, greater than mild TBI, lower extremity amputation, recent lower extremity or spine orthopedic injury requiring a profile)
2. meet criteria for moderate to severe substance-use disorder within the past month, as defined by DSM-V,
3. display behavior that would significantly interfere with validity of data collection or safety during study,
4. be in significant pain during the evaluation (7/10 by patient subjective report),
5. be a pregnant female (balance considerations), or
6. unable to communicate in English.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Across all sites, Phase One will include 50 civilians with persistent symptoms from mTBI, 50 civilian healthy controls, and 40 active duty SM healthy controls in total. Three non-military sites will test civilians. A fourth military site (FSH) will enroll and test 40 healthy active duty SMs across a range of military experience and ability levels.
  Subjects for Phase Two will include 40 active duty SMs with persistent symptoms from mTBI who are referred for physical therapy due to their symptoms. Participants will be recruited from two military medical centers specializing in the rehabilitation of active duty personnel after mTBI, WRC at Fort Carson and MAMC at Joint Base Lewis-McChord. Each site will recruit 20 participants for Aim III.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Illinois Agility Assessment | 15 minutes
  Single & dual task
Walk and Turn | 5 minutes
  Single & dual task; 1 minute long walk
Custom Turns Course | 15 minutes
  Single & dual task; walking along a marked course involving turns of varying angles
Civilian Ambulatory Task | 10 minutes
  Participants will asked to follow a series of written directions that involves walking in uncontrolled pedestrian environments. Subjects will be given a walking route through written instructions and landmark-based directions to follow. The walking route will require participants to ambulate around public areas and will take approximately 10 minutes to complete. Participants will be required to navigate through crowded hallways, ascend and descend stairs, and scan for pedestrians and/or other obstacles. The total time to complete the task will be recorded
Simulated Urban Combat Patrol | 10 minutes
  Participants will complete a simulated patrol task within a small room partitioned into two areas. Each area will contain several targets illuminated with LED lights and containing infrared (IR) sensing diodes. Participants will be instructed to enter the room, and tag all red LEDs by pointing a laser at the IR receiver located next to the LED. Participants will use a trigger-activated laser (i.e., laser gun) to tag targets. Upon being tagged with the laser, the white LEDs surrounding the target will activate to indicate the target has been cleared. The total time to complete the task will be recorded. Following the task, participants will also be asked to recount the number targets in each room.

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory | 4 minutes
  22-item patient-reported questionnaire assessing cognitive, affective, somatic, and vestibular symptoms. Total scores range: 0-88. Subscores [cognitive, affective, somatic, and vestibular] ranges: 0-22 each. The higher the value, the worse the outcome.
Dizziness Handicap Inventory | 4 minutes
  25-item patient-reported questionnaire related to dizziness, scored based on functional, emotional, and physical domains (and totaled). The higher the value, the worse the outcome. Scores range from 0 to 100 (28 possible points for physical, 36 for emotional, and 36 for functional).
Quality of Life after Brain Injury | 10 minutes
  37-item patient-reported questionnaire of health-related quality of life after a brain injury
Post-Traumatic Stress Disorder Checklist | 4 minutes
  17-item patient-reported questionnaire related to PTSD. Each item can be rated on a scale of 1 to 5. The score is totaled at the end. The higher the score, the worse the outcome. Scores range from 17 to 85
Ohio State University TBI Identification Method | 8 minutes
  A standardized procedure for determining a person's TBI history
Automated Neuropsychological Assessment Metric | 30 minutes
  A computer-based assessment of cognition
Vestibular Ocular Motor Screening | 15 minutes
  A screening tool used to detect signs and symptoms of a concussion
Revised HiMAT | 15 minutes
  A mobility assessment tool that involves various types of locomotion
Functional Gait Assessment | 15 minutes
  Assessment of postural stability during walking tasks

CONTACTS AND LOCATIONS:
Overall Officials: Laurie King, Principal Investigator — Oregon Health and Science University
Locations (6):
- United States (6):
  - Warrior Recovery Clinic, Fort Carson, Colorado
  - Courage Kenny Research Center, Minneapolis, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Fort Sam Houston, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Madigan Army Medical Center, Lakewood, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fino PC, Parrington L, Walls M, Sippel E, Hullar TE, Chesnutt JC, King LA. Abnormal Turning and Its Association with Self-Reported Symptoms in Chronic Mild Traumatic Brain Injury. J Neurotrauma. 2018 May 15;35(10):1167-1177. doi: 10.1089/neu.2017.5231. Epub 2018 Mar 23. PMID 29078732
- [Background] Scherer MR, Weightman MM, Radomski MV, Davidson LF, McCulloch KL. Returning service members to duty following mild traumatic brain injury: exploring the use of dual-task and multitask assessment methods. Phys Ther. 2013 Sep;93(9):1254-67. doi: 10.2522/ptj.20120143. Epub 2013 Jun 13. PMID 23766395
- [Background] King LA, Mancini M, Fino PC, Chesnutt J, Swanson CW, Markwardt S, Chapman JC. Sensor-Based Balance Measures Outperform Modified Balance Error Scoring System in Identifying Acute Concussion. Ann Biomed Eng. 2017 Sep;45(9):2135-2145. doi: 10.1007/s10439-017-1856-y. Epub 2017 May 24. PMID 28540448
- [Derived] Fino PC, Michielutti PG, Pelo R, Parrington L, Dibble LE, Hoppes CW, Lester ME, Weightman MM, King LA. A Hybrid Assessment of Clinical Mobility Test Items for Evaluating Individuals With Mild Traumatic Brain Injury. J Neurol Phys Ther. 2023 Apr 1;47(2):84-90. doi: 10.1097/NPT.0000000000000427. Epub 2022 Dec 19. PMID 36538333
- [Derived] Parrington L, King LA, Hoppes CW, Klaiman MJ, Michielutti P, Fino PC, Dibble LE, Lester ME, Weightman MM. Exploring Vestibular Ocular Motor Screening in Adults With Persistent Complaints After Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2022 Sep-Oct 01;37(5):E346-E354. doi: 10.1097/HTR.0000000000000762. Epub 2022 Jan 20. PMID 35067602
- [Derived] Fino PC, Weightman MM, Dibble LE, Lester ME, Hoppes CW, Parrington L, Arango J, Souvignier A, Roberts H, King LA. Objective Dual-Task Turning Measures for Return-to-Duty Assessment After Mild Traumatic Brain Injury: The ReTURN Study Protocol. Front Neurol. 2021 Jan 15;11:544812. doi: 10.3389/fneur.2020.544812. eCollection 2020. PMID 33519659